CLINICAL TRIAL: NCT05052164
Title: Improvement Of Physical And Physiological Parameters In Menopausal Or Post-Menopausal Celiac Women. Effects Of Gluten-Free Diet And Physical Exercise
Brief Title: Improvement Of Physical And Physiological Parameters In Menopausal Or Post-Menopausal Celiac Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Assistant Professor, University of Alicante
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UA-2018-10-22
Record Dates: First submitted 2021-09-07; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Celiac Disease; Diet, Gluten-Free; Exercise; Resistance Training; Quality of Life; Body Composition
MeSH Terms: conditions — Celiac Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gluten-free nutrition plan + exercise group (Experimental): Celiac women who perform a physical exercise program 3/4 times per week and a gluten-free isocaloric dietary plan.
  Interventions: Behavioral: Gluten-free nutrition plan + exercise group
- Gluten-free nutrition plan group (Experimental): Women with celiac disease following a gluten-free isocaloric dietary plan.
  Interventions: Behavioral: Gluten-free nutrition plan group
- Celiac controls group (Active Comparator): Women with celiac disease in whom all variables are measured but no intervention is performed.
  Interventions: Behavioral: Active Comparator: Celiac controls group
- Non-celiac controls group (No Intervention): Non celiac menopausal or post-menopausal in whom all the tests were measured but they did not perform an intervention program with physical exercise or special follow-up of an adapted dietary-nutritional program

INTERVENTIONS:
Behavioral: Gluten-free nutrition plan + exercise group — Menopausal or post-menopausal celiac women will follow a physical exercise program 3/4 times per week and their dietary intake will be gluten-free isocaloric
  Arms: Gluten-free nutrition plan + exercise group
Behavioral: Gluten-free nutrition plan group — Menopausal or post-menopausal celiac women will follow a gluten-free isocaloric dietary program
  Arms: Gluten-free nutrition plan group
Behavioral: Active Comparator: Celiac controls group — Menopausal or post-menopausal celiac women in whom all the tests were measured but they did not perform an intervention program with physical exercise or special follow-up of an adapted dietary-nutritional program
  Arms: Celiac controls group

SUMMARY:
Celiac disease (CD) is an immunological disorder that mainly affects the small intestine, generating an inflammatory process in response to the presence of gluten (a protein). Autoimmune diseases are part of a group of diseases that are difficult to diagnose without a specific protocol or consensus to detect them due to the number of symptoms and diseases with which it has a relationship. The incidence of CD in Spain -according to data from the rest of the European Economic Community, since there is no study on incidence in Spain- is assumed to be approximately 1 per 100 live births. It is more frequent in women, with a 2:1 ratio. The only treatment consists of a STRICT GLUTEN-FREE DIET FOR LIFE. This results in the disappearance of symptoms, normalization of serology and recovery of intestinal villi. Failure to follow the diet can lead to important complications which, especially in adulthood, can manifest themselves in the form of osteopenia, osteoporosis and a high risk of neoplasms in the digestive tract, mainly. The main objective is to achieve a physical and physiological improvement in menopausal or post-menopausal celiac women. The specific objectives will be to know the influence of a dietary-nutritional program combined with physical exercise in menopausal or post-menopausal celiac women on:

* Physical condition (strength, endurance, functional autonomy...).
* Body composition.
* Psychological aspects.
* Physiological parameters (heart rate, maximum oxygen consumption, blood analysis...).

ELIGIBILITY:
Inclusion Criteria:

* Women
* Over 40 years old
* Menopausal or post-menopausal women
* Women with celiac disease (in the case of the experimental groups)

Exclusion Criteria:

* Men
* Women of childbearing age
* Women < 40 years old
* Failure to sign informed consent form

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL) | 12 weeks
  A QoL questionnaire was performed; the WHOQOL-BREF of the World Health Organization
Body Composition - Fat Mass | 12 weeks
  Evaluation of body fat by bioimpedance.
Body Composition - Lean Body Mass | 12 weeks
  Evaluation of lean body mass by bioimpedance.
Body Composition - Visceral Fat | 12 weeks
  Evaluation of visceral fat by bioimpedance.
Weight | 12 weeks
  Weight evaluation using a digital scale
Strength | 12 weeks
  A calibrated handgrip dynamometer (Takei 5101, Tokyo, Japan) measure isometric grip strength (HGS)
Adherence to gluten-free diet | 12 weeks
  Questionnaire "Adherence to gluten-free diet" was performed.
Anthropometric assessment - Skinfolds | 12 weeks
  Restricted profile proposed by the International Society for the Development of Cineanthropometry was carried out.
Anthropometric assessment - Perimeters | 12 weeks
  Restricted profile proposed by the International Society for the Development of Cineanthropometry was carried out.
Anthropometric assessment - Diameters | 12 weeks
  Restricted profile proposed by the International Society for the Development of Cineanthropometry was carried out.
Anthropometric assessment - Height | 12 weeks
  Restricted profile proposed by the International Society for the Development of Cineanthropometry was carried out.
Resistance test | 12 weeks
  6-minute walk test. This test is an adaptation of the Rikli and Jones (1998) test.
Balance test | 12 weeks
  By means of the PSYMTEC® contact platform, which act as switches and are useful for recording contact times between supports.
Functional autonomy test | 12 weeks
  GDLAM protocol
State of mind | 12 weeks
  Evaluation by using the Profile of Mood States POMS questionnaire.
Eating disorders | 12 weeks
  Eating disorders questionnaire: Eating Attitudes Test Questionnaire (EAT) in its 26-item version (EAT-26) in Spanish (Rivas et al., 2010).
Heart rate variability | 12 weeks
  Using novel Firstbeat Bodyguard device (Föhr, 2016)
Maximum oxygen consumption | 12 weeks
  Heart rate measurement and recording with Firsbeat Bodyguard
Glucose in blood | 12 weeks
  Glucose by blood test
Cholesterol in blood | 12 weeks
  Cholesterol by blood test
Creatinine in blood | 12 weeks
  Creatinine by blood test
Urea in blood | 12 weeks
  Urea by blood test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alicante, Alicante, San Vicente Del Raspeig, Spain